CLINICAL TRIAL: NCT04215627
Title: Comparison Between Invasive Hemodynamic Monitoring, Using the PiCCO Monitor, to a Non-invasive Photoplethysmography Based Device in Hemodynamic Unstable Critically Ill Patients, With Vasopressor Support
Brief Title: Comparing the PiCCO Monitor to the Non-invasive Biobeat (BB)-316PW in ICU Patients
Status: Completed | Type: Observational
Sponsor: Biobeat Technologies Ltd. (Industry)
Collaborators: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: Biobeat004
Record Dates: First submitted 2019-12-29; First posted 2020-01-02 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Critically Ill; Hemodynamic Instability
Keywords: Critically Ill patients; blood pressure; vital signs; non-invasive monitoring; Vasopressor support
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: non-invasive monitoring — Comparing the PiCCO monitor to the non-invasive BB-613PW device in hemodynamically unstable critically ill patients in the ICU
  Other Names: BB-613PW

SUMMARY:
The aim of this study is to compare hemodynamic monitoring using the invasive PiCCO device to the BB-613PW wireless, non-invasive PPG-based device, in critically ill patients within the ICU, suffering from hemodynamic instability and in need of vasopressor support. Data will be gathered prospectively and analysed retrospectively.

ELIGIBILITY:
Inclusion Criteria:

* ICU adult patients in the need of vasopressor support of more than 0.2 mcg/Kg/Min for a period longer than 3 hours
* Patients in which PiCCO monitoring is needed

Exclusion Criteria:

* Refusal of the subject
* Technical difficulties in insertion of the PiCCO catheters
* Significant cardiac arrhythmias
* Significant valvular disease
* Pregnancy

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to the ICU unit, suffering from shock and in need for vasopressor support of more than 0.2 mcg/Kg/Min for a period longer than 3 hours, and that the treating physician has decided there is a need to insert a PiCCO catheter for invasive monitoring of their hemodynamic condition. Total period of monitoring will be up to 72 hours.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2019-12-26 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Level of accordance between the BB-613PW to the PiCCO | 72 hours per individual
  We will compare the level of accordance of blood pressure, heart rate, stroke volume, cardiac output, heart rate variability, and systemic vascular resistance.

CONTACTS AND LOCATIONS:
Overall Officials: Ayana Dvir, MD, MHA, Principal Investigator — The Assaf Harofeh Medical Center, Tzrifin, Israel
Locations (1):
- The Assaf Harofeh Medical Center, Zrifin, Rishon LeZiyyon, Israel

IPD SHARING:
Plan to Share IPD: Undecided
We plan to share the anonymised data within a manuscript (both analysed data and the raw vital sign data).